CLINICAL TRIAL: NCT02844595
Title: Behavioural Activation Treatment for Smoking Cessation and Depressive Symptomatology: a Randomized Controlled Trial
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Santiago de Compostela (Other)
Responsible Party: Principal Investigator, Elisardo Becoña Iglesias, Elisardo Becoña, University of Santiago de Compostela
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: PSI2015-66755-R (MINECO/FEDER)
Record Dates: First submitted 2016-07-19; First posted 2016-07-26 (Estimated); Last update posted 2018-10-10 (Actual); Status verified 2018-10

CONDITIONS: Smoking
Keywords: Smoking, psychological treatment, depression
MeSH Terms: conditions — Smoking; Depression

STUDY DESIGN:
Who Masked: Participant

ARMS (3):
- Standard cognitive-behavioural smoking cessation treatment (Active Comparator)
  Interventions: Behavioral: Standard cognitive-behavioural smoking cessation treatment
- Standard smoking cessation treatment and behavioral activation (Active Comparator)
  Interventions: Behavioral: Standard cognitive-behavioural smoking cessation treatment and behavioural activation
- Control group (No Intervention): It will be a delayed treatment control group for a period of 3 months.

INTERVENTIONS:
Behavioral: Standard cognitive-behavioural smoking cessation treatment — Standard cognitive-behavioural smoking cessation treatment is an effective treatment for tobacco dependence. The treatment elements are: treatment contract, self-report and graphic representation of cigarette consumption, information about tobacco, stimulus control, activities for the avoidance of withdrawal syndrome, physiological feedback (CO in expired air) on cigarette consumption, nicotine fading (change of cigarette brands each week progressively decreasing the intake of nicotine and tar), and relapse-prevention strategies (assertion training, problem solving training, change tobacco related misconceptions, management of anxiety and anger, exercise, weight control, self-reinforcing, and changing irrational beliefs).
  Treatment will be delivered in eight 60-minute sessions over 8 consecutive weeks.
  Arms: Standard cognitive-behavioural smoking cessation treatment
Behavioral: Standard cognitive-behavioural smoking cessation treatment and behavioural activation — Behavioural activation will be applied along with standard cognitive-behavioural smoking cessation treatment. The treatment elements are: those present in the standard cognitive-behavioural smoking cessation treatment, plus analysis of the relationship between behaviour and mood, identification of situations and behaviours that decrease mood, identifying avoidance behaviours, and identifying thoughts of rumination and worry, self-report of pleasant daily activities, pleasant activity scheduling to increase engagement in rewarding activities, and to reduce patterns of behavioural avoidance.
  Treatment will be delivered in eight 60-minute sessions over 8 consecutive weeks.
  Arms: Standard smoking cessation treatment and behavioral activation

SUMMARY:
The number of people who smoke, have concurrent depression and that seek treatment for smoking cessation has increased in recent years. This implies the need to design intensive and specific interventions that target this issue. In depression treatment, behavioural activation is one of the psychological interventions whose characteristics of brevity, flexibility and efficiency make it an ideal candidate to be included as part of smoking cessation treatment, especially when smokers have depressive symptoms. The aims of the present trial are: 1) to assess the efficacy (abstinence rates) of a psychological smoking cessation treatment with elements from behavioural activation for managing depressed mood (a randomized control trial with three groups: standard cognitive-behavioural smoking cessation treatment, standard cognitive-behavioural smoking cessation treatment plus behavioural activation, and a control group of delayed treatment) at the end of treatment, and at 3-, 6-, and 12-months follow-ups; and 2) to assess whether the applied cognitive-behavioural smoking cessation treatment plus behavioural activation improves depressed mood at the end of treatment and 3-, 6, 12-months follow-ups.

DETAILED DESCRIPTION:
In recent years there has been a great interest in analyzing the relationship between smoking and depression due to the high smoking rates in this population. Smokers with depression are more likely to smoke heavily, show greater tobacco dependence, suffer more severe withdrawal, experience lower quit rates and have more relapse than smokers without depression. Some studies propose the inclusion of behavioural activation techniques to standard cognitive-behavioural therapy for quitting smoking, arguing that the loss of the ability to experience pleasure in response to daily activities after quitting smoking is a significant barrier to achieving and maintaining abstinence. With this type of intervention, the exposure to positive reinforcers alternative to cigarettes increases and the resulting distress of withdrawal syndrome it is also reduced. Therefore, behavioural activation may improve smoking abstinence rates and depressive symptomatology. This project aims to assess the effectiveness of a psychological intervention for smoking cessation with components of behavioural activation for managing depressed mood. We will use a single blind controlled randomized design. Two hundred and fifty daily (≥ 10 cigarettes/day) smokers will be randomized to one of three conditions: 1) standard cognitive-behavioural smoking cessation treatment (n=100); 2) standard cognitive-behavioural smoking cessation treatment plus behavioural activation (n=100); or 3) a control group of three months delayed treatment (n=50). Both active treatments will be administered in eight weekly 60 minute sessions. The primary outcomes will be carbon monoxide (CO) verified at 24-hours point prevalence abstinence at the end of the treatment, a 7-day point prevalence abstinence at 3 months follow-up, a 30-days point prevalence abstinence at 6-, and 12-months follow-ups; and depressive symptomatology through BDI-II and Hamilton Depression Rating Scale scores at the end of treatment, and at 3-, 6-, and 12-months follow-ups. Additional aims include assessing others activation-related variables, craving, self-efficacy and withdrawal syndrome. This randomized controlled trial will be the first trial of Behavioural Activation and Smoking Cessation psychological treatment in a Spanish sample of seeking treatment smokers.

ELIGIBILITY:
Inclusion Criteria:

* 18 years of age or older who smoke at least 10 cigarettes per day
* Desire to participate voluntarily in the treatment offered to quit smoking
* Correctly fill out all the pretreatment assessment questionnaires
* Be able to provide written informed consent

Exclusion Criteria:

* To have a diagnosis of a severe mental disorder (bipolar disorder and / or psychotic disorder)
* To have a substance use disorder (alcohol, cannabis, cocaine, heroin), different from a tobacco use disorder
* To smoke rolling snuff, cigars, little cigars or other tobacco products
* To have participated in an effective psychological treatment to quit smoking during the previous 12 months
* To have received other effective pharmacological treatment to quit smoking in the previous 12 months (nicotine gum or patches, bupropion, varenicline)
* To have a physical pathology involving life threatening risks for the person who would require immediate intervention in individual format (eg. Recent myocardial infarction, pneumothorax, etc.)

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 275 (Actual)
Dates: Start 2016-01; Primary Completion 2018-06 (Actual); Study Completion 2018-06 (Actual)

PRIMARY OUTCOMES:
Point-prevalence abstinence | 1 year
  Participants will be considered abstinent if they report abstinence, not even a puff of a cigarette, for ≥24 hours at the end of treatment (week 8 since beginning treatment), and for ≥7 days prior to follow up day at 3 months follow-up and have an expired carbon monoxide reading of ≤10 parts per million. At 6-, and 12-months follow-ups, participants will be considered abstinent if they report abstinence, not even a puff of a cigarette, for ≥30 days prior to follow up day and have an expired carbon monoxide reading of ≤10 parts per million.
Change from baseline in depressive symptoms on the Beck Depression Inventory-II (BDI-II) | 1 year
Change from baseline in depressive symptoms on the Hamilton Depression Rating Scale | 1 year

SECONDARY OUTCOMES:
Continuous abstinence | 1 year
  According to the Russell Standard (West et al., 2005), participants will be considered abstinent if they report abstinence, have smoke not more than five cigarettes from the start of the abstinence period, and have an expired carbon monoxide reading of ≤10 parts per million
Reduction of cigarette consumption | 1 year
  Reduction of cigarette consumption by 50% or more between baseline and each follow-up will be calculated from the number of cigarettes smoked in the past 7 days at the end of treatment (week 8 since beginning treatment) and at 3 months follow-up. At 6-, and 12-months follow-ups it will be calculated from the number of cigarettes smoked in the past 30 days.
Change from baseline in the Environmental Reward Observation Scale (EROS) scores | 1 year
Change from baseline in the Behavioural Activation for Depression Scale (BADS) scores | 1 year

CONTACTS AND LOCATIONS:
Overall Officials: Elisardo Becoña, Principal Investigator — University of Santiago de Compostela
Locations (1):
- Smoking Cessation and Addictive Disorders Unit, Faculty of Psychology, University of Santiago de Compostela, Santiago de Compostela, A Coruña, Spain

REFERENCES:
- [Background] Cook JW, Piper ME, Leventhal AM, Schlam TR, Fiore MC, Baker TB. Anhedonia as a component of the tobacco withdrawal syndrome. J Abnorm Psychol. 2015 Feb;124(1):215-25. doi: 10.1037/abn0000016. Epub 2014 Nov 10. PMID 25384069
- [Background] Gierisch JM, Bastian LA, Calhoun PS, McDuffie JR, Williams JW Jr. Smoking cessation interventions for patients with depression: a systematic review and meta-analysis. J Gen Intern Med. 2012 Mar;27(3):351-60. doi: 10.1007/s11606-011-1915-2. Epub 2011 Oct 26. PMID 22038468
- [Background] Hitsman B, Papandonatos GD, McChargue DE, DeMott A, Herrera MJ, Spring B, Borrelli B, Niaura R. Past major depression and smoking cessation outcome: a systematic review and meta-analysis update. Addiction. 2013 Feb;108(2):294-306. doi: 10.1111/add.12009. PMID 23072580
- [Background] MacPherson L, Tull MT, Matusiewicz AK, Rodman S, Strong DR, Kahler CW, Hopko DR, Zvolensky MJ, Brown RA, Lejuez CW. Randomized controlled trial of behavioral activation smoking cessation treatment for smokers with elevated depressive symptoms. J Consult Clin Psychol. 2010 Feb;78(1):55-61. doi: 10.1037/a0017939. PMID 20099950
- [Derived] Theodoulou A, Fanshawe TR, Leavens E, Theodoulou E, Wu AD, Heath L, Stewart C, Nollen N, Ahluwalia JS, Butler AR, Hajizadeh A, Thomas J, Lindson N, Hartmann-Boyce J. Differences in the effectiveness of individual-level smoking cessation interventions by socioeconomic status. Cochrane Database Syst Rev. 2025 Jan 27;1(1):CD015120. doi: 10.1002/14651858.CD015120.pub2. PMID 39868569
- [Derived] Lopez-Duran A, Martinez-Vispo C, Barroso-Hurtado M, Suarez-Castro D, Becona E. Incorporating technology in smoking cessation interventions: In-person vs. Video-call formats. Int J Med Inform. 2025 Mar;195:105774. doi: 10.1016/j.ijmedinf.2024.105774. Epub 2024 Dec 24. PMID 39742855
- [Derived] Martinez-Vispo C, Rodriguez-Cano R, Lopez-Duran A, Senra C, Fernandez Del Rio E, Becona E. Cognitive-behavioral treatment with behavioral activation for smoking cessation: Randomized controlled trial. PLoS One. 2019 Apr 8;14(4):e0214252. doi: 10.1371/journal.pone.0214252. eCollection 2019. PMID 30958831
- [Derived] Becona E, Martinez-Vispo C, Senra C, Lopez-Duran A, Rodriguez-Cano R, Fernandez Del Rio E. Cognitive-behavioral treatment with behavioral activation for smokers with depressive symptomatology: study protocol of a randomized controlled trial. BMC Psychiatry. 2017 Apr 8;17(1):134. doi: 10.1186/s12888-017-1301-7. PMID 28390417